CLINICAL TRIAL: NCT02763462
Title: The Etiology of Acute Febrile Illness Requiring Hospitalization (AFIRE). A Multicenter Study of the Indonesia Research Partnership on Infectious Disease (INA-RESPOND)
Brief Title: The Etiology of Acute Febrile Illness Requiring Hospitalization
Acronym: AFIRE
Status: Completed | Type: Observational
Sponsor: Ina-Respond (Other)
Collaborators: National Institute of Health Research and Development, Ministry of Health Republic of Indonesia (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: INA101; U1111-1263-2248 (Other: WHO UTN Number); HHSN261200800001E (Other: NIAID); HHSN261201500003I (Other: NIAID)
Record Dates: First submitted 2016-04-04; First posted 2016-05-05 (Estimated); Results first posted 2023-02-27 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Acute Febrile Illness
Keywords: Acute Febrile Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, buffy coat, urine, throat swab, nasal swab.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is an observational cohort study of hospitalized patients with fever. This study will collect demographic data, history of illness, signs and symptoms, results of laboratory tests, clinical course, treatment and outcome. This study conducted at eight INA-RESPOND hospitals. Potential study patients will be any patients (both children and adults).

DETAILED DESCRIPTION:
This study is an observational cohort to identify the etiologies of acute febrile illness (less than or equal to 2 weeks), which are thought to be endemic or novel in a certain area. Therefore, there are no hypotheses that require sample size calculation to be tested. It is expected that this study will enroll a minimum of 200 patients per site: approximately 100 adults and 100 pediatric cases. The final sample size is therefore estimated to be 1600.

Primary Objective:

To identify the etiology of acute febrile illness cases and evaluate clinical manifestations and outcomes.

Secondary Objectives:

1. To provide clinical data that are essential for improving and/or developing clinical management and health policies.
2. To enhance research capacity and networking for infectious diseases in Indonesia by improving clinical research site capability in conducting research relevant to public health.
3. To establish a repository of biological specimens for future study, such as determining the etiology of undiagnosed fever and/or its pathogenicity and its public health importance.

This study will be conducted at all the INA-RESPOND hospitals (8 hospitals):

* Dr. Cipto Mangunkusumo Hospital , Jakarta
* Penyakit Infeksi Prof. Dr. Sulianti Saroso Hospital, Jakarta
* Dr. Hasan Sadikin Hospital, Bandung
* Dr. Kariadi Hospital, Semarang
* Dr. Sardjito Hospital, Yogyakarta
* Dr. Soetomo Hospital, Surabaya
* Sanglah Hospital, Bali
* Dr. Wahidin Soedirohusodo Hospital, Makassar

The study will enroll eligible fever patients for a period of up to 1 year. Follow-up may be up until one year after last subject is enrolled. Stored samples will be investigated during the study and/or after study completion.

After enrollment, patients will be seen at 14-28 days and at 3 months post enrollment. Patients will be seen every 3 months (6, 9, and 12 months within a window period of +/- 14 days) until cured and no related symptoms persists or the one year time point is reached. The samples will be collected for storage at enrollment, the 14-28 day visit, at 3 months and every 3 months thereafter if not cured.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥1 year
* Acute febrile illness requiring hospitalization (fever defined as temperature recorded ≥38.0°C during the first 24 hour period of hospitalization).
* Hospitalized within the past 24 hours.
* Willing to allow storage of blood and other specimens for use in future studies of infectious diseases.

Exclusion Criteria:

* Hospitalized within the past 3 months, not including current hospitalization for acute febrile illness.
* Inpatient transfer from another hospital.
* A known medical disorder or other circumstance, which in the opinion of the PI might make the participation of the individual unsafe or difficult.

Examples include, but not limited to: mental illness which could affect compliance with protocol, an anemic patient preventing blood draw.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with acute febrile illness.
Sampling Method: Probability Sample
Enrollment: 1492 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. dr. M. Hussein Gasem, PhD, SpPD-KPTI, Principal Investigator — University of Diponegoro/ Dr. Kariadi hospital; Prof. Emiliana Tjitra, MSC, Ph.D, Principal Investigator — NIHRD, Indonesia; Dr. Bachti Alisjahbana, PhD, SpPD-KPTI, Principal Investigator — Univerversity of Padjajaran / Dr. Hasan Sadikin Hospital
Locations (8):
- Indonesia (8):
  - University of Udayana/Sanglah Hospital, Denpasar, Bali
  - University of Diponegoro/ Dr. Kariadi Hospital, Semarang, Central Java
  - University of Indonesia/ Dr. Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta
  - Penyakit Infeksi Sulianti Saroso Hospital, Jakarta, DKI Jakarta
  - University of Airlangga/ Dr. Soetomo Hospital, Surabaya, East Java
  - University of Padjajaran/ Dr. Hasan Sadikin Hospital, Bandung, West Java
  - University of Hassanudin/ Dr. Wahidin Sudirohusodo Hospital, Makassar
  - University of Gadjah Mada/ Dr. Sardjito Hospital, Yogyakarta

IPD SHARING:
Plan to Share IPD: No
No plan to share data

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was done from July 2013 until October 2016
Pre-assignment Details: From total target 1600 subjects only achieved 1492 subjects enrolled.
Groups:
- Hospitalized Participants With Acute Febrile Illness.: Hospitalized patients with any infectious diseases with cardinal symptoms at acute fever (<= 2 weeks)
Period: Overall Study
Arm/Group | Hospitalized Participants With Acute Febrile Illness.
Started | 1492
Completed | 1486
Not Completed | 6
Not completed — Protocol Violation | 6

BASELINE CHARACTERISTICS:
Population: We analyzed all subjects enrolled and excluded 6 participants who were not eligible.
Groups:
- Hospitalized Participants With Acute Febrile Illness: Hospitalized patients with any infectious disease with cardinal symptoms of acute fever (<= 2 weeks).
Arm/Group | Hospitalized Participants With Acute Febrile Illness
Number analyzed (Participants) | 1486
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 623
  Between 18 and 65 years | 793
  >=65 years | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.6 (19.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 656
  Male | 830
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1486
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1486
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Indonesia | 1486

OUTCOME MEASURES:

1. Primary Outcome: The Etiologies (Bacteria, Viruses, Parasites, Fungi and Others) of Fever Illness Expressed in Percentages of Enrolled Subjects.
Description: Any pathogens identified as a caused of febrile illness based on laboratory tests such as blood culture, other culture (sputum/ pus/ urine/ feces), serology, and molecular.
Time Frame: Total length of time the subject will be in the study is 3 months after enrollment or until cured or maximum 1 year.
Population: All participants who have specimens to be tested
Measure: Count of Participants; unit: Participants
Groups:
- Hospitalized Participants With Acute Febrile Illness: Hospitalized patients with any infectious disease with cardinal symptoms of acute fever (<=2 weeks)
Arm/Group | Hospitalized Participants With Acute Febrile Illness
Number analyzed (Participants) | 1486
Participants
  Viruses | 621
  Bacteria | 362
  Parasites | 15
  Multiple pathogens | 5
  Unidentified pathogens | 483

2. Secondary Outcome: Number of Participants With Affected Organ System by Each Specific Pathogen
Description: The organ system affected induced clinical symptoms that provide essential information for improving clinical management in differentiating between each identified pathogen.
Time Frame: 3 years
Population: The organ system affected induced clinical symptoms that provide essential information for improving clinical management in differentiating between each identified pathogen.
Measure: Number; unit: participants
Groups:
- Central Nervous System; Upper Respiratory; Lower Respiratory; Skin and Soft Tissue; Gastrointestinal; Genitourinary; Constitutional; Multiorgan: Organ system affected based on identified pathogens.
Arm/Group | Central Nervous System | Upper Respiratory | Lower Respiratory | Skin and Soft Tissue | Gastrointestinal | Genitourinary | Constitutional | Multiorgan
Number analyzed (Participants) | 9 | 22 | 43 | 20 | 378 | 1 | 41 | 489
participants
  Dengue | 4 | 7 | 0 | 8 | 226 | 1 | 27 | 194
  Salmonella spp. | 1 | 3 | 1 | 0 | 37 | 0 | 5 | 56
  Rickettsia spp. | 0 | 0 | 1 | 3 | 48 | 0 | 6 | 45
  Influenza | 1 | 4 | 10 | 0 | 4 | 0 | 0 | 49
  Leptospira spp. | 0 | 1 | 0 | 0 | 19 | 0 | 0 | 24
  Chikungunya | 1 | 1 | 1 | 1 | 10 | 0 | 2 | 21
  E.Coli | 0 | 1 | 2 | 0 | 9 | 0 | 0 | 9
  S. pneumoniae | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 17
  M. tuberculosis | 0 | 2 | 5 | 0 | 1 | 0 | 0 | 12
  Multiple pathogens | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
  Other single pathogen | 1 | 2 | 22 | 7 | 23 | 0 | 1 | 59

3. Secondary Outcome: Number of Participants Enrolled Per Each Clinical Research Site
Description: Eight clinical research sites in 7 cities in Indonesia have been established to conduct clinical research that improved research capacity and networking for Infectious diseases in Indonesia.
Time Frame: 3 years
Population: Eight clinical research sites in 7 cities in Indonesia have been established to conduct clinical research that improved research capacity and networking for Infectious diseases in Indonesia.
Measure: Count of Participants; unit: Participants
Groups:
- Number of Subject Enrolled: Number of subject enrolled per each clinical research sites.
Arm/Group | Number of Subject Enrolled
Number analyzed (Participants) | 1486
Participants
  RSUP dr Hasan Sadikin | 269
  RSUP Sanglah | 213
  RSUPN Dr Cipto Mangunkusumo | 65
  RSPI Prof Dr Sulianti Saroso | 91
  RSUP dr Wahidin Sudirohusodo | 201
  RSUP dr Kariadi | 257
  RSUD dr Soetomo | 221
  RSUP dr Sardjito | 169

4. Secondary Outcome: Number of Vials Stored Based on Specimen Type
Description: Each clinical research site and reference laboratory have been established to have capability to store repository specimen for future study.
Time Frame: 3 years
Population: Each clinical research site and reference laboratory have been established to have capability to store repository specimen for future study.
Measure: Number; unit: vials
Units Other Than Participants: vials
Groups:
- Number of Specimens Stored.: Number of specimens stored based on specimen type.
Arm/Group | Number of Specimens Stored.
Number analyzed (Participants) | 14099
Number analyzed (vials) | 14099
vials
  Plasma EDTA | 7032
  Buffy coat | 2311
  Sputum | 29
  Pleural fluid | 2
  Feces | 27
  Nasopharyngeal swab | 114
  Urine | 205
  LCS | 4
  Pus | 4
  DNA | 2487
  RNA | 1884

ADVERSE EVENTS:
Time Frame: 48 hours after study related blood drawn
Description: Any untoward or unfavorable medical occurrence in a human subject that occurs within 48 hours of a study-related blood draw that is possibly, probably, or definitely related to the blood draw. Any event outside of this 48 hour window period will not be considered an AE for this study.
Arm/Group | Hospitalized Participants With Acute Febrile Illness
All-Cause Mortality (participants affected / at risk) | 89/1486
Serious Adverse Events (participants affected / at risk) | 0/1486
Other Adverse Events (participants affected / at risk) | 8/1486
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hospitalized Participants With Acute Febrile Illness (N=1486)
Hematoma (Skin and subcutaneous tissue disorders) | 6 (7) — Hematoma at the site where blood is drawn
Fever (General disorders) | 1 (1) — Fever, chills, sweating
Convulsion (Nervous system disorders) | 1 (1) — Convulsion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No